CLINICAL TRIAL: NCT05295901
Title: The Effect of the Mobile Application Developed to Provide Symptom Control in Chronic Obstructive Pulmonary Patients on Self-Efficacy and Chronic Disease Management
Brief Title: The Effect of Mobile Health Applications on Symptom Control, Self-efficacy and Chronic Disease Management in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Neşe Özdemir, research assistant, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COPD And Mobile Application
Record Dates: First submitted 2022-01-22; First posted 2022-03-25 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: copd; chronic disease; mobile healthy applications
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Intervention Model Description: randomized controlled quasi-experimental study
Who Masked: Participant
Masking Description: participants do not know that they are in the experimental or control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the pre-test phase (first interview) - Patient Diagnosis Form, COPD Self-efficacy Scale, Chronic Disease Care Assessment Scale-Patient Form, COPD Assessment Test (CAT), Modified Medical Research Council (mMRC) Dyspnea Scale average 15-20 min. will be implemented.
  After the pre-test, the mCOPD mobile application will be installed on the phones of the patients and it will be checked whether the mobile application is working. mobile application content will be explained. In addition, a pulse oximeter device will be given to the patients by the researcher to record their pulse and saturation values and its use will be explained.
  In the final test phase (final interview); The COPD Self-Efficacy Scale, the Chronic Disease Care Assessment Scale-Patient Form, the COPD Assessment Test (CAT), the Modified Medical Research Council (mMRC) Dyspnea Scale and the Satisfaction Questionnaire will be applied to determine the degree of satisfaction
  Interventions: Device: mKOAH application
- control group (No Intervention): In the pre-test phase (first interview); Patient Diagnosis Form, COPD self-efficacy scale, Chronic Disease Care Assessment Scale-Patient Form, COPD Assessment Test (CAT), Modified Medical Research Council (MRC) Dyspnea Scale will be applied. No action will be taken after the interview.
  In the final testing phase (final interview); After applying the COPD Self-Efficacy Scale, the Chronic Disease Care Assessment Scale-Patient Form, the COPD Assessment Test (CAT), the Modified Medical Research Council (MRC) Dyspnea Scale, the mCOPD application will be installed on their phones and training

INTERVENTIONS:
Device: mKOAH application — mobile app installed group
  Arms: experimental group

SUMMARY:
Name:The effect of the mobile application developed to provide symptom control in chronic obstructive pulmonary patients on self-efficacy and chronic disease management

Aim:Considering the covid-19 pandemic seen all over the world, it is aimed to develop a mobile application with an integrated care model that allows individuals with chronic obstructive pulmonary disease to control their symptoms that seriously affect their quality of life.

DETAILED DESCRIPTION:
In recent years, mobile technologies have been used in the use of self-management applications. Mobile technologies have the opportunity to provide information exchange between the patient and the healthcare professional, to provide patient-specific personalized training, to provide reminders, warnings reinforcements, to increase motivation and behavior change, Reducing the impact of exacerbations through early recognition of symptoms and prompt treatment of individuals with COPD has been shown to be effective in reducing the risk of hospitalization, improving health-related quality of life, and controlling the burden of COPD.In addition, due to the COVID-19 pandemic experienced all around the world, telehealth and mobile technologies were used in the delivery of health services in many countries.

Importance of Research

Considering the covid-19 pandemic seen all over the world and in our country aim to develop a mobile application, which is an integrated care model that allows individuals with chronic obstructive pulmonary disease to control their symptoms that seriously affect their quality of life.

Method

Data Collection Tools

1. Patient Diagnosis Form: The "Patient Diagnosis Form", prepared by the researcher in line with the literature, consists of two parts.

   Section 1: Age, place of residence, gender, educational status, occupation, economic status, health insurance, living with whom, smoking and alcohol consumption status, cigarette pack years, COPD information source, etc. for the patient. will consist of questions.

   Section 2: COPD diagnosis, presence of other diseases, number of symptoms and attacks, medication used, etc. questions were included
2. COPD Self-Efficacy Scale) (CSES):The scale consists of 34 items that determine the degree of self-confidence of COPD patients to manage or avoid breathing difficulties during certain activities, and five sub-dimensions: negative impact, emotional state, physical effort, weather/environment influence, and behavioral risk factors.
3. Chronic Disease Care Assessment Scale-Patient Form:The Likert-type and 20-item scale consists of five sub-dimensions: patient participation, decision making, goal setting, problem solving, and monitoring/coordination
4. COPD Assessment Test (CAT):It is a scale consisting of 8 parameters in which the effects of the disease on daily life and health status are determined.
5. Modifiye Medical Research Council (mMRC)/ Dyspnea Scale:It was used to compare the severity of dyspnea during activity in people with and without lung disease.
6. Satisfaction Form: It is a form scored from 1 to 5 by the researcher in order to determine how satisfied the experimental group is with the content of the application at the end of the study.
7. mCOPD mobile app:The conceptual and theoretical framework of the mobile application designed for individuals with COPD has been developed based on the chronic care model.Inside the mKOAH mobile application; There are interfaces under the headings of education, management, evaluation, vital parameters, communication, about us, resources.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Having and using a smartphone (Android or iPhone)
* who have been diagnosed with COPD
* no communication problem
* Not having mental confusion or any psychiatric problems
* Individuals who agree to participate in Stage 2 (50%≤FEV1<80) and Stage 3 (30%≤FEV1<50) and Stage 4 (FEV1<30) research who meet the GOLD 2021 criteria will be included in the study.

Exclusion Criteria:

* with cognitive dysfunction
* Comorbid diseases such as severe pulmonary, cardiological and malignant disease
* in exacerbation
* Visual, hearing, cognitive, or dexterity impairment that precludes mobile use
* Patients in Stage 1 (FEV1≥80%) meeting the GOLD 2021 criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Application of the patient diagnosis form before the intervention was made to the experimental group | 1 months
  Patient Diagnosis Form: Prepared by the researcher in line with the literature, consists of two parts.
  Section 1: Age, place of residence, gender, educational status, occupation, economic status, health insurance, living with whom, smoking and alcohol consumption status, cigarette pack years, COPD information source, etc. for the patient. will consist of questions.
  Section 2: COPD diagnosis, presence of other diseases, number of symptoms and attacks, medication used, etc. questions were included
Application of the COPD self-efficacy scale to the experimental group before the intervention | 1 months
  COPD Self-Efficacy Scale (CSES):The scale consists of 34 items that determine the degree of self-confidence of COPD patients to manage or avoid breathing difficulties during certain activities, five sub-dimensions: negative impact, emotional state, physical effort, weather/environment influence behavioral risk factors. High scores on managing or avoiding breathing difficulties interpreted as an increase in the degree of confidence.
Application of the patient form scale to evaluate the chronic disease care before the intervention to the experimental group | 1 months
  Chronic Disease Care Assessment Scale-Patient Form:The Likert-type and 20-item scale consists of five sub-dimensions: patient participation, decision making, goal setting, problem solving, and monitoring/coordination. An increase in the scale score indicates that individuals with chronic diseases are satisfied with the care they receive and that chronic disease management is sufficient.
Application of the pre-intervention COPD assessment scale to the experimental group | 1 months
  COPD Assessment Test (CAT):It is a scale consisting of 8 parameters in which the effects of the disease on daily life and health status are determined.The scores of the questions in the test vary between "0-40". The CAT evaluation test score is 0-10 "low impact", 11-20 "medium impact", 21-30 "high impact", and 31-40 " very high impact" evaluated as .
Application of the dyspnea scale to the experimental group before the intervention | 1 months
  Modifiye Medical Research Council (mMRC)/ Dyspnea Scale:It was used to compare the severity of dyspnea during activity in people with and without lung disease. Scoring is between 0-4. Above 1 point indicates severe respiratory distress.
Application of the patient diagnosis form to the control group | 1 months
  Patient Diagnosis Form: Prepared by the researcher in line with the literature, consists of two parts.
  Section 1: Age, place of residence, gender, educational status, occupation, economic status, health insurance, living with whom, smoking and alcohol consumption status, cigarette pack years, COPD information source, etc. for the patient. will consist of questions.
  Section 2: COPD diagnosis, presence of other diseases, number of symptoms and attacks, medication used, etc. questions were included
Application of the COPD self-efficacy scale to the control group | 1 months
  COPD Self-Efficacy Scale (CSES):The scale consists of 34 items that determine the degree of self-confidence of COPD patients to manage or avoid breathing difficulties during certain activities, five sub-dimensions: negative impact, emotional state, physical effort, weather/environment influence behavioral risk factors. High scores on managing or avoiding breathing difficulties interpreted as an increase in the degree of confidence.
Application of the chronic disease care assessment scale to the control group | 1 months
  Chronic Disease Care Assessment Scale-Patient Form:The Likert-type and 20-item scale consists of five sub-dimensions: patient participation, decision making, goal setting, problem solving, and monitoring/coordination.An increase in scale scores indicates that individuals with chronic disease are satisfied with the care they receive and that chronic disease management is sufficient.
Application of the COPD assessment scale to the control group | 1 months
  COPD Assessment Test (CAT):It is a scale consisting of 8 parameters in which the effects of the disease on daily life and health status are determined.The scores of the questions in the test vary between "0-40". The CAT evaluation test score is 0-10 "low impact", 11-20 "medium impact", 21-30 "high impact", and 31-40 "very high impact" evaluated as .
Application of the dyspnea scale to the control group | 1 months
  Modifiye Medical Research Council (mMRC)/ Dyspnea Scale:It was used to compare the severity of dyspnea during activity in people with and without lung disease.Scoring is between 0-4. Above 1 point indicates severe respiratory distress.

SECONDARY OUTCOMES:
application of the COPD self-efficacy scale to the experimental group after the intervention | 3 months
  COPD Self-Efficacy Scale (CSES):The scale consists of 34 items that determine the degree of self-confidence of COPD patients to manage or avoid breathing difficulties during certain activities, five sub-dimensions: negative impact, emotional state, physical effort, weather/environment influence behavioral risk factors. High scores on managing or avoiding breathing difficulties interpreted as an increase in the degree of confidence.
Application of the patient form to evaluate the chronic disease care after the intervention in the experimental group | 3 months
  Chronic Disease Care Assessment Scale-Patient Form:The Likert-type and 20-item scale consists of five sub-dimensions: patient participation, decision making, goal setting, problem solving, and monitoring/coordination.An increase in scale scores indicates that individuals with chronic disease are satisfied with the care they receive and that chronic disease management is sufficient.
Application of the COPD assessment scale to the experimental group after the intervention | 3 months
  COPD Assessment Test (CAT):It is a scale consisting of 8 parameters in which the effects of the disease on daily life and health status are determined.The scores of the questions in the test vary between "0-40". The CAT evaluation test score is 0-10 "low impact", 11-20 "medium impact", 21-30 "high impact", and 31-40 "high impact" evaluated as .
Application of the dyspnea scale to the experimental group after the intervention | 3 months
  Modifiye Medical Research Council (mMRC)/ Dyspnea Scale:It was used to compare the severity of dyspnea during activity in people with and without lung disease.Scoring is between 0-4. Above 1 point indicates severe respiratory distress.
Application of the post-intervention satisfaction form to the experimental group | 3 months
  Satisfaction Form: It is a form scored from 1 to 5 by the researcher in order to determine how satisfied the experimental group is with the content of the application at the end of the study.
Application of the COPD self-efficacy scale to the control group | 3 months
  COPD Self-Efficacy Scale (CSES):The scale consists of 34 items that determine the degree of self-confidence of COPD patients to manage or avoid breathing difficulties during certain activities, five sub-dimensions: negative impact, emotional state, physical effort, weather/environment influence behavioral risk factors. High scores on managing or avoiding breathing difficulties interpreted as an increase in the degree of confidence.
Application of the chronic disease care assessment scale to the control group | 3 months
  Chronic Disease Care Assessment Scale-Patient Form:The Likert-type and 20-item scale consists of five sub-dimensions: patient participation, decision making, goal setting, problem solving, and monitoring/coordination.An increase in scale scores indicates that individuals with chronic disease are satisfied with the care they receive and that chronic disease management is sufficient.
Application of the COPD assessment scale to the control group | 3 months
  COPD Assessment Test (CAT):It is a scale consisting of 8 parameters in which the effects of the disease on daily life and health status are determined.The scores of the questions in the test vary between "0-40". The CAT evaluation test score is 0-10 "low impact", 11-20 "medium impact", 21-30 "high impact", and 31-40 "very high impact" evaluated as .
Application of the dyspnea scale to the control group | 3 months
  Modifiye Medical Research Council (mMRC)/ Dyspnea Scale:It was used to compare the severity of dyspnea during activity in people with and without lung disease.Scoring is between 0-4. Above 1 point indicates severe respiratory distress.

CONTACTS AND LOCATIONS:
Overall Officials: Neşe ÖZDEMİR, PhD student, Principal Investigator — Muş Alparslan University
Locations (1):
- Neşe ÖZDEMİR, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta N, Agrawal S, Chakrabarti S, Ish P. COPD 2020 Guidelines - what is new and why? Adv Respir Med. 2020;88(1):38-40. doi: 10.5603/ARM.2020.0080. No abstract available. PMID 32153009
- [Background] Halpin DMG, Celli BR, Criner GJ, Frith P, Lopez Varela MV, Salvi S, Vogelmeier CF, Chen R, Mortimer K, Montes de Oca M, Aisanov Z, Obaseki D, Decker R, Agusti A. The GOLD Summit on chronic obstructive pulmonary disease in low- and middle-income countries. Int J Tuberc Lung Dis. 2019 Nov 1;23(11):1131-1141. doi: 10.5588/ijtld.19.0397. PMID 31718748
- [Background] Bernard S, Boucher S, McLean L, Moffet H. Mobile technologies for the conservative self-management of urinary incontinence: a systematic scoping review. Int Urogynecol J. 2020 Jun;31(6):1163-1174. doi: 10.1007/s00192-019-04012-w. Epub 2019 Jul 2. PMID 31267139
- [Background] Baker E, Fatoye F. Patient perceived impact of nurse-led self-management interventions for COPD: A systematic review of qualitative research. Int J Nurs Stud. 2019 Mar;91:22-34. doi: 10.1016/j.ijnurstu.2018.12.004. Epub 2018 Dec 31. PMID 30669076
- [Background] Alghamdi SM, Rajah AMA, Aldabayan YS, Aldhahir AM, Alqahtani JS, Alzahrani AA. Chronic Obstructive Pulmonary Disease Patients' Acceptance in E-Health Clinical Trials. Int J Environ Res Public Health. 2021 May 14;18(10):5230. doi: 10.3390/ijerph18105230. PMID 34069028